CLINICAL TRIAL: NCT07028749
Title: Phase 2b Randomized, Double-Blind, Parallel-Group, Placebo-Controlled Study of MAR001 in Patients With Elevated Triglycerides and Remnant Cholesterol (TYDAL-TIMI 78)
Brief Title: Study of MAR001 in Adults With Elevated Triglycerides and Remnant Cholesterol
Acronym: TYDAL-TIMI 78
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Marea Therapeutics (Industry)
Collaborators: The TIMI Study Group (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MAR-103
Record Dates: First submitted 2025-06-11; First posted 2025-06-19 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Hypertriglyceridemia
Keywords: Hypertriglyceridemia; MAR001; Remnant Cholesterol; TYDAL; TIMI-78
MeSH Terms: conditions — Hypertriglyceridemia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- MAR001 Dose 1 (Experimental): Subcutaneous injection
  Interventions: Drug: MAR001; Drug: Placebo
- MAR001 Dose 2 (Experimental): Subcutaneous Injection
  Interventions: Drug: MAR001; Drug: Placebo
- MAR001 Dose 3 (Experimental): Subcutaneous Injection
  Interventions: Drug: MAR001; Drug: Placebo

INTERVENTIONS:
Drug: MAR001 — Subcutaneous Injection
Drug: Placebo — Subcutaneous injection

SUMMARY:
The primary objective of the study is to evaluate the effect of MAR001 compared to placebo on levels of the TG and RC in adults with elevated TG and RC.

ELIGIBILITY:
Inclusion Criteria:

* Elevated fasting TGs and RC
* Elevated nonfasting TGs and RC
* Fasting LDL-C ≥ 50 mg/dL (≥ 1.29 mmol/L) and ≤ 130 mg/dL (≤ 3.36 mmol/L)
* Willingness to provide informed consent and comply with the intervention and all study assessments
* Stable diet for a minimum of 3 months prior to screening and with no plans to change diet through duration of study
* Stable drug regimen (if relevant) prior to screening visit and no planned changes during screening or trial participation

Exclusion Criteria:

* Acute or chronic liver disease
* TG concentration ≥880mg/dl
* History of type 1 diabetes mellitus or history of diabetic ketoacidosis
* Newly diagnosed T2DM
* Participants with known active hepatitis A, B, or C
* Uncontrolled hypothyroidism
* Any condition that prevents the participant from complying with study procedures

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 216 (Estimated)
Dates: Start 2025-06-30 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Primary Endpoint | 12 weeks
  Change from baseline in fasting TG compared to placebo. Change from baseline in fasting RC compared to placebo.

SECONDARY OUTCOMES:
Secondary Endpoint | 12 weeks
  Change in fasting VLDL-C Change in fasting non-HDL-C MAR001 Concentrations over time

CONTACTS AND LOCATIONS:
Locations (54):
- United States (26):
  - Marea Site 328, Anniston, Alabama
  - Marea Site 329, Mobile, Alabama
  - Marea Site 313, Little Rock, Arkansas
  - Marea Site 306, Hamden, Connecticut
  - Marea Site 302, Boca Raton, Florida
  - Marea Site 307, Port Saint Lucie, Florida
  - Marea Site 310, Columbus, Georgia
  - Marea Site 319, Peachtree Corners, Georgia
  - Marea Site 317, Park Ridge, Illinois
  - Marea Site 325, Springfield, Illinois
  - Marea Site 301, Louisville, Kentucky
  - Marea Site 316, Baltimore, Maryland
  - Marea Site 330, Kansas City, Missouri
  - Marea Site 305, St Louis, Missouri
  - Marea Site 304, Great Neck, New York
  - Marea Site 318, New Windsor, New York
  - Marea Site 303, Greensboro, North Carolina
  - Marea Site 315, Winston-Salem, North Carolina
  - Marea Site 314, Greenville, South Carolina
  - Marea Site 320, Little River, South Carolina
  - Marea Site 326, Memphis, Tennessee
  - Marea Site 322, Amarillo, Texas
  - Marea Site 308, McKinney, Texas
  - Marea Site 312, San Antonio, Texas
  - Marea Site 321, Manassas, Virginia
  - Marea Site 309, Tacoma, Washington
- Australia (13):
  - Marea Site 103, Canberra, Australian Capital Territory
  - Marea Site 105, Kanwal, New South Wales
  - Marea Site 107, Merewether, New South Wales
  - Marea Site 106, Miranda, New South Wales
  - Marea Site 109, Wollongong, New South Wales
  - Marea Site 108, Herston, Queensland
  - Marea Site 104, Milton, Queensland
  - Marea Site 111, Leabrook, South Australia
  - Marea Site 102, Clayton, Victoria
  - Marea Site 110, Heidelberg Heights, Victoria
  - Marea Site 113, Hoppers Crossing, Victoria
  - Marea Site 101, Nedlands, Western Australia
  - Marea Site 112, Perth, Western Australia
- Canada (7):
  - Marea Site 406, Concord, Ontario
  - Marea Site 403, London, Ontario
  - Marea Site 404, Sarnia, Ontario
  - Marea Site 401, Chicoutimi, Quebec
  - Marea Site 402, Montreal, Quebec
  - Marea Site 405, Québec, Quebec
  - Marea Site 407, Québec, Quebec
- New Zealand (8):
  - Marea Site 211, Birkenhead, Auckland
  - Marea Site 207, New Lynn, Auckland
  - Marea Site 203, Papatoetoe, Auckland
  - Marea Site 205, Silverdale, Auckland
  - Marea Site 206, Christchurch, South Island
  - Marea Site 204, Ebdentown, Upper Hutt
  - Marea Site 209, Christchurch
  - Marea Site 208, Rotorua

IPD SHARING:
Plan to Share IPD: Undecided